CLINICAL TRIAL: NCT04869852
Title: Effects of Mango Intake on Skin Health and Gut Microbiome Changes in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MANGO_02
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Photoaging
Keywords: Wrinkles; Polyphenols; Vitamins
MeSH Terms: interventions — Food

STUDY DESIGN:
Intervention Model Description: Healthy postmenopausal women aged 50 - 70, Fitzpatrick skin type I, II, or III
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango (Experimental): 85g mango, 4x/week
  Interventions: Other: Food
- No Mango (No Intervention): No mango intake

INTERVENTIONS:
Other: Food — 85g mango, 4x/week
  Arms: Mango

SUMMARY:
Mangos are a rich source of nutrients such as carotenoids, vitamin C and fiber, as well as polyphenols and phenolic acids such as mangiferin, ellagic acid, and gallotannins. Mango extract has been reported to protect against photo-aging of the skin in an animal model exposed to UVB radiation, reducing the length of wrinkles and increasing collagen bundles. Beta-carotene and other carotenoids are known to provide skin protection from sunlight, but other compounds in mangos, may also be important in reducing oxidative damage in aging skin.

We have recently completed a pilot study showing a clear trend in skin wrinkle reduction when postmenopausal women consumed 85g of Ataulfo mangos, four times per week for 16 weeks. To confirm and extend these results, a larger study is proposed.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 70 years old
* Postmenopausal
* Fitzpatrick skin type I, II, or III
* BMI 18.5 - 35
* Must be willing to comply with all protocol requirements
* Must be willing to have flash photo facial images taken with the imaging systems

Exclusion Criteria:

* Smokers
* Allergy to mangos
* Vegans/vegetarians
* Adults unable to consent

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Wrinkles | week 20
  Wrinkle score measured by Facial Image Analysis System

SECONDARY OUTCOMES:
Facial Hydration | week 20
  Moisture measured by MoistureMeterSC
Facial Redness | week 20
  Redness measured by Facial Image Analysis System
Facial Elasticity | week 20
  measured by Cutometer
Gut microbiome | week 20
  analyze for changes in gut microbiome diversity measures (Shannon Diversity)
Gut microbiome | week 20
  Analyze for the relative abundance of short chain fatty acid producing bacteria

IPD SHARING:
Plan to Share IPD: No